CLINICAL TRIAL: NCT05103111
Title: Effect of Forward Head Posture on Temporomandibular Joint Proprioception in Postmenopausal Women. an Observational Study
Brief Title: Effect of FHP on TMJ Proprioception in Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, manal ahmed el-shafei mohamed, lecturer of physical therapy for women's health, Cairo University
Other Study IDs: P.T.REC/012/003297
Record Dates: First submitted 2021-09-28; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FHP group (study group): it will be consisted of 50 women, suffering from FHP (CVA is less than 48°)
  Interventions: Other: No intervention
- control group (without FHP): it will be consisted of 50 women, not having FHP (CVA is more than 48°).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no intervention

SUMMARY:
anterior protrusion of head in relation to the trunk; It has a high prevalence among old women as increased age is associated with a reduced cervical range of motion (ROM), greater thoracic kyphosis which is associated with greater cervical flexion and greater forward head posture accompanying with greater deficits in cervical ROM of flexion and rotation. So, the aim of the study is to determine the effect of forward head posture on temporomandibular joint proprioception in postmenopausal women

DETAILED DESCRIPTION:
A convenient sample of 100 postmenopausal women will be participated in this study; they are divided into 2 groups according to their cranio-vertebral angle (CVA). The FHP group will be consisted of 50 women, suffer from FHP (CVA was less than 48°). The control group will be consisted of 50 women, are free from FHP (CVA more than 48°).

The participants will be recruited from Faculty of Physical Therapy, Cairo University and Faculty of Physical Therapy, MUST University. Informed consent will be obtained from each participant after explaining the nature, purpose, and benefits of the study, informing them of their right to refuse or withdraw at any time, and about the confidentiality of any obtained information.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* their age will range from 50 to 60 years
* their body mass index (BMI) will range from 25 to 28 kg/m2

Exclusion Criteria:

* any identified or acquired dental defects
* existing dental prosthesis use, visual, voice and hearing disabilities
* facial paralysis
* orofacial, neck or shoulder fractures or procedures
* fixed or mobile spinal deformity
* headache
* migraine
* any vestibular or neurological condition that may impair TMJ proprioception.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The postmenopausal women will be divided into two groups according to their cranio-vertebral angle (CVA). The FHP group will consist of 50 women, suffering from FHP (CVA is less than 48°). The control group will consist of 50 women, not having FHP (CVA is more than 48°).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-03-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of cranio-vertebral angle (CVA) | up to 3 months
  The CVA is angle formed by a horizontal line drawn through the spinous process of seventh cervical vertebra c7 and line connecting spinous process of c7 and tragus of the ear. the markers will be placed on c7 and tragus of the ear and a photo will be captured by using digital camera from lateral view for three times .Then, the photographs of the woman are then transferred to the device to be analyzed by the Surgimap spine programme which by measuring the angle between a horizontal line passing through C7 and a line extending from the tragus of the ear to C7, calculated the positions of the anatomical points on the photographs to calculate the CVA ,the average of 3 times measurement will be taken, the cut-off point for CVA was 48 °; the woman with less than 48 ° CVA is considered having FHP, whereas the woman with more than 48 ° CVA is considered healthy .
Measurement of mouth opening angle | up to 3 months
  The woman will be instructed to open her mouth as much as possible. The calliper then calculated the vertical distance between the incisal edge of the maxillary central incisor and the labioincisal edge of the opposing mandibular incisor.
Measurement of mandibular protrusion | up to 3 months
  The initial position was the physiological resting position (average space of 3 mm between the occlusal surfaces of the maxillary and mandibular teeth) of the mandible . The woman was told from that role to shift her mandible anteriorly without contact with the tooth. The calliper then measured the gap from the incisal edge of the maxillary central incisor to the incisal edge of the mandibular central incisor.
Measurement of lateral movements of the mandible | up to 3 months
  The initial position was the physiological resting position from which the woman was advised to shift her mandible to the right and then to the left as far as possible. Then the calliper assessed the distance between the labioincisal embrasures of the maxillary central incisor to the labioincisal embrasure of the opposing mandibular incisor.Then, to measure the functional ROM of TMJ, the full ROM of TMJ in each direction was divided by three. In each direction, the caliper was adjusted at the functional ROM to train the woman to move her jaw from the starting position to that functional ROM for 3 times. Then for 3 times with open eyes and 3 times with closed eyes, the woman was asked to shift her jaw actively from the star-ting position to the functional ROM of each direction and the therapist assessed the ROM by the digital caliper in each time.

CONTACTS AND LOCATIONS:
Overall Officials: Manal Ahmed, lecturer, Principal Investigator — lecturer of physical therapy for women's health, Cairo university

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF